CLINICAL TRIAL: NCT02537379
Title: A Prospective Observational Post-Marketing Study of Sovaldi® Plus Copegus® in Japanese Patients With Chronic Genotype 2 Hepatitis C Virus Infection
Brief Title: Use-Results Surveillance Study of Sovaldi® Plus Copegus® in Japanese Patients With Chronic Genotype 2 Hepatitis C Virus Infection
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-334-1444 / COPE1501
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C virus; observational; post-marketing; sofosbuvir
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; Ribavirin

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SOF+COPE: Adult patients with genotype 2 chronic HCV infection with or without compensated cirrhosis who take SOF+COPE as part of routine clinical care at a participating clinical site.
  Interventions: Drug: SOF; Drug: COPE

INTERVENTIONS:
Drug: SOF — SOF 400 mg tablets administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: COPE — COPE tablets administered orally in a divided daily weight-based dose according to the package insert for the approved Copegus® labeling in Japan (< 60 kg = 600 mg , > 60 kg to ≤ 80 kg = 800 mg, and > 80 kg = 1000 mg)
  Other Names: Copegus®; Ribavirin

SUMMARY:
This post-marketing surveillance (PMS) study for Sovaldi® tablets (sofosbuvir, SOF) administered in combination with Copegus® tablets (ribavirin, COPE) will evaluate the safety and efficacy of SOF administered in combination with ribavirin under real world use in Japan. Among adult patients with chronic genotype 2 hepatitis C virus (HCV) infection and treated with SOF+ribavirin in routine clinical use, the primary objective of this study is to evaluate the incidence of adverse drug reactions (ADRs) under real world settings.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult patients with serogroup 2 (genotype 2) chronic HCV infection with or without compensated cirrhosis
* Patients who are prescribed SOF+COPE

Key Exclusion Criteria:

* None

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with serogroup 2 (genotype 2) chronic HCV infection with or without compensated cirrhosis who take SOF+COPE as part of routine clinical care at a participating clinical site.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reaction (ADR) under real world settings | Up to 16 weeks

SECONDARY OUTCOMES:
Proportion of participants with sustained virologic response (SVR) 12 and 24 weeks after discontinuation of therapy (SVR12 and SVR24) | Posttreatment Weeks 12 and 24
  SVR12 and SVR24 are defined as HCV RNA < the lower limit of quantification (LLOQ) 12 and 24 weeks following the last dose of study drug, respectively.
Proportion of participants with HCV NS5B resistance associated variants among patients who do not achieve SVR at 12 weeks | Approximately 12 weeks after treatment completion or discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (45):
- Japan (45):
  - Amagasaki-shi
  - Asahi-shi
  - Asahikawa-shi
  - Beppu-shi
  - Chichibu-shi
  - Fujioka-shi
  - Fukui-shi
  - Hamamatsu
  - Iizuka-shi
  - Inzai-shi
  - Ishinomaki-shi
  - Iwaki
  - Izunokuni-shi
  - Kahoku-gun
  - Kanazawa
  - Kirishima-shi
  - Kisarazu-shi
  - Kitamoto-shi
  - Kobe
  - Koshigaya-shi
  - Kure-shi
  - Moriguchi-shi
  - Nagakute-shi
  - Nagaoka-shi
  - Nagasaki
  - Nagoya
  - Nakagami-gun
  - Nanto-shi
  - Nishinomiya-shi
  - Ofukeshi
  - Okayama
  - Ome-shi
  - Osaka
  - Ōta-ku
  - Sapporo
  - Sasebo-Shi
  - Sendai
  - Shinagawa-ku
  - Shinjuku-ku
  - Tokorozawa-shi
  - Tokushima
  - Wakayama
  - Yachiyo-shi
  - Yokohama
  - Yufu-shi